CLINICAL TRIAL: NCT07275073
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, Immunogenicity, and Preliminary Antitumor Activity of JMT106 Injection in Patients With Advanced Solid Tumors
Brief Title: JMT106 Injection in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMT106-001
Record Dates: First submitted 2025-08-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor; Lung Squamous Cell Carcinoma; Hepatocellular Carcinoma
Keywords: solid tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JMT106 injection as single agent (Experimental)
  Interventions: Drug: JMT106 Injection

INTERVENTIONS:
Drug: JMT106 Injection — Use according to the protocol.

SUMMARY:
This study is the first-in-human Phase I study of JMT106 injection, comprising two phases: Dose escalation with backfill and cohort expansion. The planned study population consists of subjects with advanced solid tumors. The objective is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of JMT106 injection as monotherapy in participants with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically confirmed advanced solid tumor.
3. Failure of at least one line of standard therapy, or no standard treatment available, or intolerant to standard treatment at the current stage.
4. At least one measurable lesion according to RECIST 1.1 criteria.
5. ECOG performance status of 0-1.
6. Expected survival ≥3 months.
7. Sufficient organ function, with laboratory tests meeting the following criteria (no blood transfusion or hematopoietic growth factor treatment within 14 days):

   1. Absolute neutrophil count (ANC) ≥1.5×10⁹/L;
   2. Platelets (PLT) ≥90×10⁹/L;
   3. Hemoglobin (Hb) ≥90 g/L;
   4. Total bilirubin (TBIL) ≤1.5×ULN (≤3×ULN for liver metastases or hepatocellular carcinoma);
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN for liver metastases or hepatocellular carcinoma);
   6. Creatinine clearance (Ccr) >50 mL/min (calculated by Cockcroft-Gault formula);
   7. Activated partial thromboplastin time (APTT) ≤1.5×ULN; INR ≤1.5×ULN.
8. Fertile participants (male and female) must agree to use reliable contraception (hormonal, barrier, or abstinence) with their partners during the trial and for at least 180 days after the last dose. Female participants of childbearing potential must have a negative blood pregnancy test within 7 days before enrollment.
9. Understand and voluntarily sign the informed consent form (ICF).

Exclusion Criteria:

1. Previous treatment with anti-GPC3 therapy.
2. Presence of spinal cord compression or clinically active central nervous system metastases (untreated or symptomatic metastases, or those requiring corticosteroids/anticonvulsants for symptom control), or carcinomatous meningitis. Patients with previously treated brain metastases (e.g., whole-brain radiotherapy or stereotactic brain radiotherapy) may be enrolled if clinically stable for ≥4 weeks with no imaging evidence of progressive brain metastases.
3. Long-term immunosuppressive therapy (e.g., cyclosporine) or daily systemic steroid therapy (e.g., >20 mg prednisone or equivalent), excluding those using nasal spray, inhaled, or other topical glucocorticoid therapies.
4. Adverse reactions from prior antitumor therapy not recovered to CTCAE 5.0 Grade ≤1 (excluding toxicities deemed non-risky by the investigator, e.g., alopecia).
5. Any antitumor therapy (chemotherapy, targeted therapy, immunotherapy, etc.) or investigational intervention within 4 weeks or 5 half-lives (whichever is shorter) before the first dose, or traditional Chinese medicine with antitumor indications within 14 days prior.
6. Grade ≥3 immune-related adverse events (irAEs, per CTCAE 5.0) from prior immunotherapy.
7. Concurrent participation in another interventional clinical trial (observational trials or follow-up phases allowed).
8. Major surgery within 28 days before the first dose or planned tumor resection during the study.
9. Significant bleeding tendency within 4 weeks before the first dose, or high-risk conditions (e.g., gastrointestinal hemorrhage, severe hemoptysis) per investigator judgment; hereditary bleeding disorders.
10. Known severe allergy to the study drug or its excipients.
11. Active bacterial, fungal, or viral infection requiring IV treatment within 14 days before randomization (prophylactic therapy allowed if no active infection symptoms); patients with viral hepatitis are allowed to receive antiviral treatment.
12. Uncontrolled effusions (pleural, peritoneal, pericardial) requiring frequent drainage or intervention within 14 days before the first dose (excluding cytologic evaluation of effusions).
13. History of allogeneic organ or hematopoietic stem cell transplantation.
14. Immunodeficiency, including HIV-positive status.
15. HBsAg-positive or HBcAb-positive with HBV-DNA >2000 IU/mL; HCV antibody-positive with HCV-RNA positivity.
16. History of tuberculosis treatment within 2 years before the first dose.
17. Interstitial lung disease or severe pulmonary dysfunction.
18. History of inflammatory bowel disease or chronic diarrhea.
19. Severe cardiovascular/cerebrovascular disease, including:

    1. Severe arrhythmias/conduction abnormalities (e.g., ventricular arrhythmias requiring intervention, AV block grade II-III);
    2. Acute coronary syndrome, congestive heart failure, stroke, or other Grade ≥3 cardiovascular events within 6 months before the first dose;
    3. NYHA class ≥II or LVEF <50%;
    4. Long QTc syndrome or QTc >480 ms (Fridericia formula), or concomitant use of QTc-prolonging drugs;
    5. Uncontrolled hypertension (systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg at screening).
20. Other active malignancies within 2 years (except cured localized tumors, e.g., basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer, in situ prostate/cervical/breast cancer).
21. Live vaccination within 28 days before the first dose (inactivated vaccines, e.g., seasonal flu vaccine, allowed).
22. Pregnancy or lactation.
23. Other conditions deemed unsuitable by the investigator (e.g., depression history/current treatment, psychiatric disorders affecting compliance, main portal vein tumor thrombus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE), | Up to 2 years
  Assess the incidence of all AE and serious adverse events (SAE)..
Maximum Tolerated Dose (MTD), | Up to 1 years
  MTD is defined as the dose level at which the estimated value of toxicity probability is closest to the target toxicity rate (i.e., 0.3).
Dose-Limiting Toxicity (DLT) | Up to 1 years
  Evaluate the incidence of DLT in different dose groups.
Dose for Expansion (RDE) | Up to 1 years
  Explore the recommended dose for the cohort expansion phase.
Recommended Phase 2 Dose (RP2D) | Up to 1 years
  Recommended phase II dose
Overall Response Rate (ORR) | ORR as Assessed by Investigator according to RECIST v1.1
  Up to 2 years

SECONDARY OUTCOMES:
Plasma concentrations and pharmacokinetic (PK) parameters | About 6 months after first dosing
  Tests are conducted after administration of JMT106.
2. Title: ORR | Up to 2 years
  ORR as Assessed by Investigator according to RECIST v1.1
Disease Control Rate (DCR) | Up to 2 years
  DCR according to RECIST v1.1
Progression-Free Survival (PFS) | Up to 2 years
  PFS as Determined by Investigator according to RECIST v1.1
Duration of Response (DoR) | Up to 2 years
  DOR as Assessed by Investigator according to RECIST v1.1
Incidence and titers of anti-drug antibodies (ADAs) to JMT106, and incidence of neutralizing antibodies (NAbs, if applicable) | About 6 months after first dosing
  Tests are conducted after administration of JMT106.
Plasma concentrations of JMT106 | About 6 months after first dosing
  Tests are conducted after administration of JMT106.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affilicated Hospital,Zhejiang University School of Medicine, Zhejiang, China